CLINICAL TRIAL: NCT06949878
Title: Clinical Evaluation of Different Concentrations of Hydrochloric Acid Based as Micro Abrasive Kits in Management of Patients With Mild to Moderate Fluorosis (A 6month Randomized Clinical Trial)
Brief Title: 21% Hydrochloric Acid Based Versus 6.6 % Hydrochloric Based Micro Abrasive Kit in Management of Patients With Mild to Moderate Fluorosis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yaqeen Atef AbdelRazeq Mohammed, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Opertive 4
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Enamel Discoloration; Fluorosis, Dental
Keywords: Dental fluorosis; Microabrasion; Enamel Discoloration; Patient Reported Outcome Measures; Randomized clinical trial; High consentration hydrochloric acid based microabrasive kit(Antivet); Low consentration hydrochloric acid based microabrasive kit ( opalustre)
MeSH Terms: conditions — Fluorosis, Dental | interventions — opalustre

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antivet (Experimental): Complete stain removal from the Enamel Use a compact cotton swab (3 mm) to apply Antivet solution (Dental Continental, México)to the stained dental piece according to manufacturer's instructions.
  Replace the swab as it becomes stained and continue until the stain is removed. " This may take 1-5 minutes per tooth, but do not exceed 15 minutes in total. " We will keep the tooth moist during the process for effective results and avoid reusing stained cotton swab.
  Then we will apply the neutralizing solution to the tooth with a brush or micro brush, ensuring it reaches the gingival margin. Leave it on for 2 minutes.
  Once the antivet solution is neutralized, rinse the area and remove the rubber dam.
  Interventions: Drug: Antivet
- :opalustre (Experimental): Complete stain removal from the Enamel. Product will be applied to the surface with a 1 mm thick layer; ten applications of 60s to help penetration of the gel into the enamel.
  Using an abrasive rubber cup (OpalCup™ Ultradent) in contra-angle low-speed handpiece at low revolution.
  Then will be rinsed with injectable water for 30 seconds between each application
  Interventions: Drug: opalustre

INTERVENTIONS:
Drug: Antivet — Complete stain removal from the Enamel-Use a compact cotton swab (3 mm) to apply Antivet solution (Dental Continental, México)to the stained dental piece according to manufacturer's instructions.-Replace the swab as it becomes stained and continue until the stain is removed. " This may take 1-5 minutes per tooth, but do not exceed 15 minutes in total. " - We will keep the tooth moist during the process for effective results and avoid reusing stained cotton swab.-Then we will apply the neutralizing solution to the tooth with a brush or micro brush, ensuring it reaches the gingival margin. Leave it on for 2 minutes.-Once the antivet solution is neutralized, rinse the area and remove the rubber dam.
  Arms: Antivet
Drug: opalustre — Complete stain removal from the Enamel. Product will be applied to the surface with a 1 mm thick layer; ten applications of 60s to help penetration of the gel into the enamel.- Using an abrasive rubber cup (OpalCup™ Ultradent) in contra-angle low-speed handpiece at low revolution.- Then will be rinsed with injectable water for 30 seconds between each application.
  Arms: :opalustre

SUMMARY:
compare the clinical performance of different concentrations of hydrochloric acid based as micro abrasive kits in management of patients with mild to moderate fluorosis over 6month follow up .

DETAILED DESCRIPTION:
microabrasion is a permanent cosmetic dentistry treatment indeed to preserve the health of all part of any defect in enamel.

ELIGIBILITY:
Inclusion Criteria:

Patients who wanted to change the appearance of their stained teeth Males or females. Patients with three or more stained incisors and canines Patients willing and able to attend periodic follow-up visits Patient concerning with oral health. Co-operative patients who show interest to participate in the study.

Exclusion Criteria:

Patients with known allergic or adverse reaction to the tested materials. Smoking habit Patients having Poor oral hygiene Patients with special health care needs or any systemic disease that may affect treatment Patients participating in other dental studies. Patients suffering from white spot lesion, hypoplasia, amelogenesis imperfecta, dentinogenesis imperfecta, or badly broken and missing teeth due to MIH.

Participants who had a history of dental bleaching.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of treatment success | T( Time ) T0(base line )=Immediately , T1 = 3 Months , T2 = 6 Month
  Enamel discoloration or texture by Spectrophotometer Vita EasyShade When totally removed of fluorotic white spots = success & when stains doesn't removed and surface irregular = failure

SECONDARY OUTCOMES:
Clinical evaluation of Sensitivity | Time frame : T( Time ) T0(base line )=Immediately , T1 = 3 Months , T2 = 6 Month
  Patient reported outcome measures by visual analog scale (VAS) Is used to describe sensitivity by patient themselves in scores as ( o : no sensitivity) ( 10 : highly sensitive )
Patient satisfaction with the Treatment. | Time frame : T( Time ) T0(base line )=Immediately , T1 = 3 Months , T2 = 6 Month
  Patient reported outcome measures by 4-point Likert scale used to describe patient satisfaction with treatment as [(a) "yes, very satisfied", (b) "yes, mostly satisfied", (c) "less satisfied", (d) "not at all satisfied"].

IPD SHARING:
Plan to Share IPD: Yes